CLINICAL TRIAL: NCT02009943
Title: A Randomized Pilot Study of Ferric Carboxymaltose as Compared to Iron Sucrose for the Treatment of Functional Iron Deficiency Associated With Surgical Critical Illness
Brief Title: Randomized Study Comparing Ferric Carboxymaltose to Iron Sucrose to Treat Fe Deficiency in the Surgically Critically Ill
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Inadequate funds
Sponsor: Denver Health and Hospital Authority (Other)
Responsible Party: Principal Investigator, Fredric Pieracci, Assistant Professor of Surgery, Denver Health and Hospital Authority
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: COMIRB 13-3151
Record Dates: First submitted 2013-12-05; First posted 2013-12-12 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: ICU Anemia; Functional Iron Deficiency
Keywords: critical illness; iron supplementation; functional iron deficiency; ICU anemia; red blood cell transfusion
MeSH Terms: conditions — Critical Illness | interventions — ferric carboxymaltose; Ferric Oxide, Saccharated

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Ferric carboxymaltose (FDA IND pending) (Experimental): 15 mg/kg, up to 750 mg IV x 1 on the day of study enrollment.
  Interventions: Drug: Ferric carboxymaltose
- Iron sucrose (FDA IND 109,877) (Active Comparator): Iron sucrose 100 mg IV will be dosed daily using goal-direction up to a total of 700 mg over a 7-day period. Specifically, iron sucrose will be dosed daily if:
  1. TSAT < 25%
  2. Serum iron concentration < 150 ug/mL
  3. Serum ferritin concentration < 1,500 ng/mL
  Interventions: Drug: Iron sucrose
- Control (No Intervention): No iron supplementation

INTERVENTIONS:
Drug: Ferric carboxymaltose — One time dosing
  Other Names: Injectafer
  Arms: Ferric carboxymaltose (FDA IND pending)
Drug: Iron sucrose — Goal-directed dosing
  Arms: Iron sucrose (FDA IND 109,877)

SUMMARY:
Critically ill surgical patients are observed to have a functional iron deficiency which contributes to anemia, iron-deficient erythropoiesis, and an increased red blood cell transfusion requirement. Previously, iron supplementation has been studied in this population with the administration of enteral ferrous sulfate and intravenous iron sucrose but without robust results in resolving serum and bone marrow iron debts.

Ferric carboxymaltose (FCM) is novel iron-containing complex that allows for the administration of a large dose of iron over a short infusion period to allow for sustained delivery of iron to target tissues with minimal hypersensitivity reactions. While there has been reported increased efficacy and comparable safety of FCM when compared to iron sucrose in the outpatient setting, there is no data comparing these two medications in surgical critical illness.

The aim of this pilot trial is to compare two novel dosing schemes of these medications for treatment of functional iron deficiency in surgical ICU patients. The investigators hypothesize that iron supplementation with FCM, as compared to both iron sucrose and placebo, is more effective and equally safe for replacing the serum iron debt.

DETAILED DESCRIPTION:
The inflammatory response associated with surgical critical illness rapidly induces a functional iron deficiency, characterized by hypoferremia, decreased transferrin saturation (TSAT), hyperferritinemia, and iron-deficient erythropoiesis (IDE). This functional iron deficiency both contributes to intensive care unit (ICU) anemia and increases the packed red blood cell (pRBCs) transfusion requirement.

The goals of iron supplementation of critically ill surgical patients are to reverse the serum iron debt, eliminate IDE, improve anemia, and decrease pRBCs transfusions. Issues surrounding iron supplementation of this patient population include formulation, dose, route of administration, and mitigation of the complications of iron overload, including infection.

The investigators first randomized clinical trial (RCT) of iron supplementation of critically ill surgical patients compared enteral ferrous sulfate 325 mg thrice daily to placebo (NCT00450177). Although a significant reduction in pRBCs transfusion requirement for the iron group was observed, low injury severity, intolerance of enteral medications, and a predominance of traumatic brain injury limited generalizability. In a second multicenter RCT, the investigators compared intravenous iron sucrose 100 mg thrice weekly to placebo among critically ill trauma patients (NCT01180894). Iron supplementation at this dose increased the TSAT only marginally (and not above the normal range) and increased the serum ferritin concentration significantly; however, there was no effect on IDE, anemia, or pRBCs transfusion requirement. In no instance did iron supplementation increase the risk of infection, despite a relatively high incidence of marked hyperferritinemia (serum ferritin concentration > 1,000 ng/mL) in the iron group.

The severity of both the serum and bone marrow iron debts observed in these trials led us to investigate alternative dosing schemes that deliver larger quantities of bioavailable iron safely. Ferric carboxymaltose (FCM) is a novel iron-containing complex that allows for the administration of a large replenishment dose of iron (up to 750 mg) over a short infusion period. Several pharmacodynamic properties of FCM render it appealing for use in the treatment of functional iron deficiency associated with surgical critical illness, including a short infusion time, a controlled, sustained delivery of iron to target tissues over a relatively long period of time (up to one week), and minimal hypersensitivity reactions. Increased efficacy and comparable safety have been reported for FCM as compared to iron sucrose for treatment of outpatients with iron-deficiency anemia. There are currently no data regarding the efficacy of FCM for the indication of functional iron deficiency associated with surgical critical illness.

The aim of the current pilot trial is to compare two novel dosing schemes for treatment of functional iron deficiency in surgical ICU patients, both of which involve delivery of a larger total dose of iron as compared to both NCT00450177 and NCT01180894. The investigators hypothesize that iron supplementation with FCM, as compared to both iron sucrose and placebo, is more effective and equally safe for replacing the serum iron debt.

ELIGIBILITY:
Inclusion Criteria:

* Anemia (hemoglobin < 12 g/dL).
* Functional iron deficiency:

  1. Serum iron concentration < 40 ug/dL
  2. TSAT < 25%
  3. Serum ferritin concentration > 28 ng/mL
* < 72 hours from ICU admission.
* Expected ICU length of stay ≥ 7 days.

Exclusion Criteria:

* Age < 18 years.
* Active bleeding requiring pRBCs transfusion
* Iron overload (serum ferritin concentration ≥ 1,500 ng/mL). The serum ferritin concentration is an acute phase reactant that is increased during critical illness regardless of total body iron [3]. Substantial levels of hyperferritinemia (serum ferrinin concentration > 1,000 ng/dL) were observed in both NCT00450177 and NCT01180894 without increased risk of infection and despite both low TSAT and IDE. For these reasons, we believe that relative hyperferritinemia (serum ferritin concentration 500 - 1,500 ng/dL) is neither harmful nor indicative of bone marrow iron availability.
* Infection, defined using US Centers for Disease Control and Prevention (CDC) guidelines, with the exception of ventilator-associated pneumonia (VAP), which is defined as clinical suspicion for pneumonia along with a lower respiratory tract culture with ≥ 105 colony forming units per mL.
* Chronic inflammatory conditions (e.g., systemic lupus erythematosis, rheumatoid arthritis, ankylosing spondilitis).
* Pre-existing hematologic disorders (e.g., thalassemia, sickle cell disease, hemophilia, von Willibrand's disease, or myeloproliferative disease).
* Macrocytic anemia (admission mean corpuscular volume ≥ 100 fL).
* Current or recent (within 30 days) use of immunosuppressive agents.
* Use of any recombinant human erythropoietin formulation within the previous 30 days.
* Pregnancy or lactation.
* Legal arrest or incarceration.
* Prohibition of pRBCs transfusion.
* Stay of ≥ 48 hours duration in the ICU of a transferring hospital.
* History of intolerance or hypersensitivity to iron.
* Moribund state in which death was imminent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-02 (Estimated); Primary Completion 2017-08 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Reversal of the serum iron debt as measured by the transferrin saturation | One week
  Because only a small fraction of total body iron is dissolved in blood, the TSAT is currently regarded as the most accurate indicator of iron substrate available for deposition in the bone marrow and eventual incorporation into erythrocytes. Data from outpatients indicate that TSAT is a more reliable predictor of hemoglobin response as compared to either serum iron concentration or serum ferritin concentration, with a target TSAT of 25-50% considered ideal for bone marrow iron delivery. In NCT01180894, TSAT began and remained <16% despite iron supplementation with iron sucrose 100 mg IV thrice weekly. The target TSAT for this trial will be 25%-50%.

SECONDARY OUTCOMES:
Bone marrow iron debt | One week
  Bone marrow iron debt as measured by daily erythrocyte zinc protoporphyrin (eZPP) concentration. During normal erythropoiesis, iron is chelated to protoporphyrin IX to form heme. When inadequate iron is delivered to the bone marrow, zinc is substituted for iron, forming zinc protoporphyrin. An elevated eZPP is diagnostic of IDE and reflects the bone marrow iron supply regardless of total body iron.
Serum ferritin concentration | One week
  The amount of ferritin in whole blood, measured in nanograms per deciliter
Hemoglobin | 28 days
  The amount of hemoglobin in whole blood, measured in grams per deciliter
Red blood cell transfusion requirement | 28 days
  Total number of units transfused.
Nosocomial infections | 28 days
  Infections will be defined according to the US CDC guidelines, with the exception of ventilator-associated pneumonia (VAP), which is defined as clinical suspicion for pneumonia along with a lower respiratory tract culture with ≥ 105 colony forming units per mL.

CONTACTS AND LOCATIONS:
Overall Officials: Fredric M Pieracci, MD, MPH, Principal Investigator — Denver Health and Hospital
Locations (1):
- Denver Health Medical Center, Denver, Colorado, United States